CLINICAL TRIAL: NCT00687505
Title: A Phase 1, Open-Label, Dose-Finding Study Evaluating the Safety and Pharmacokinetics of FP-1039 in Subjects With Metastatic or Locally Advanced Unresectable Solid Tumors
Brief Title: Safety Study of FP-1039 To Treat Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Five Prime Therapeutics, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP1039-001
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — FP-1039

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Single ascending doses
  Interventions: Drug: FP-1039

INTERVENTIONS:
Drug: FP-1039 — Intravenous weekly administration

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of FP-1039, a new biologic treatment for cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with metastatic or locally advanced unresectable solid tumors for which standard curative or supportive measures do not exist or are no longer effective
* Male or female 18 years of age or older

Exclusion Criteria:

* Presence or history of melanoma
* Primary brain tumor
* Presence or history of glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Karmanos Cancer Institute, Detroit, Michigan
  - START (South Texas Accelerated Research Therapeutics), San Antonio, Texas